CLINICAL TRIAL: NCT03913104
Title: Feasibility and Acceptability of Dispensing Mifepristone Via Mail Order Pharmacy
Brief Title: Mail Order Mifepristone Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daniel Grossman, MD (Other)
Responsible Party: Sponsor-Investigator, Daniel Grossman, MD, Professor and Director of ANSIRH, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-26819
Record Dates: First submitted 2019-04-03; First posted 2019-04-12 (Actual); Results first posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-07

CONDITIONS: Abortion Early; Pregnancy Related
MeSH Terms: interventions — Mifepristone

STUDY DESIGN:
Intervention Model Description: Prospective Cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Medication Abortion Patients (Experimental): Oral Mifepristone 200 mg, followed by misoprostol 800 mcg administered buccally (at 24-48 hours following mifepristone)
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Mifepristone — Patients will have MifeprexⓇ (mifepristone) shipped to a preferred address via an online mail order pharmacy rather than standard care at clinic visit.

SUMMARY:
This study aims to evaluate the feasibility, acceptability, and effectiveness of dispensing mifepristone via a mail-order pharmacy. The investigators will recruit patients at up to 10 primary care and internal medicines sites not currently providing abortion services around the country, as well as abortion clinic sites. Patients will go through routine in clinic visits to determine eligibility and then will receive the medications in the mail at their preferred address. The investigators will survey patients 3 and 14 days after the initial clinic visit and interview providers at the end of the study.

DETAILED DESCRIPTION:
This is a prospective cohort study of patients obtaining medication abortion via mifepristone dispensed from an online mail order pharmacy. After an initial pilot test with 25 patients, the investigators will identify 10 clinics to participate in the study. The study team will train primary care providers not currently providing abortion to provide medication abortion with the medications dispensed via mail order pharmacy. The investigators aim to recruit up to 650 patients for this study across all the sites. Patients will come in for an initial consult visit at the study site and then receive their medications at a preferred address within 3 days of the initial visit. Study participants will fill out surveys about their experience and feedback about the acceptability of the process; this will occur at 3 and 14 days after the initial recruitment visit. The investigators will also collect clinic data from patients and clinic sites to track clinical outcomes. And the investigators will interview providers at the end of the study to better understand their experiences prescribing mifepristone via mail-order.

ELIGIBILITY:
Inclusion Criteria:

* Women seeking medication abortion through 63 days gestation
* Eligible for MifeprexⓇ at a study site
* English or Spanish speaking
* Willing and able to participate in the study, including willing and able to receive medications at home or other preferred address within 3 days of initial medication abortion visit

Exclusion Criteria:

* Not pregnant
* Not seeking medication abortion
* under the age of 15
* Over 63 days gestation
* Contraindicated for medication abortion

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 536 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Grossman, MD, Principal Investigator — University of California, San Francisco
Locations (11):
- United States (11):
  - Highland Hospital, Oakland, California
  - Children's Hospital Oakland, Oakland, California
  - Planned Parenthood Rocky Mountains, Denver, Colorado
  - Christiana Care Health System, Wilmington, Delaware
  - Atlanta Comprehensive Wellness Clinic, Atlanta, Georgia
  - Albert Einstein College of Medicine, New York, New York
  - Southern Tier Women's Health Services, Vestal, New York
  - Delaware County Women's Center, Chester, Pennsylvania
  - Allegheny Reproductive Health Center, Pittsburgh, Pennsylvania
  - Brown Family Medicine, Pawtucket, Rhode Island
  - Lifespan, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raifman S, Gurazada T, Beaman J, Biggs MA, Schwarz EB, Gold M, Grossman D. Primary care and abortion provider perspectives on mail-order medication abortion: a qualitative study. BMC Womens Health. 2024 Jul 3;24(1):382. doi: 10.1186/s12905-024-03202-z. PMID 38956609
- [Derived] Grossman D, Raifman S, Morris N, Arena A, Bachrach L, Beaman J, Biggs MA, Hannum C, Ho S, Schwarz EB, Gold M. Mail-order pharmacy dispensing of mifepristone for medication abortion after in-person clinical assessment. Contraception. 2022 Mar;107:36-41. doi: 10.1016/j.contraception.2021.09.008. Epub 2021 Sep 20. PMID 34555420

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 536 patients were consented and enrolled as part of this study. Four participants enrolled twice and were analyzed based on their abortion instance, leading to 540 abortions analyzed as part of this study.
Units Other Than Participants: Number of abortions
Period: Overall Study
Arm/Group | Medication Abortion Patients
Started | 536; 540 Number of abortions
Patient's Clinical Outcome Information Obtained | 506; 510 Number of abortions
Completed | 506; 510 Number of abortions
Not Completed | 30; 30 Number of abortions
Not completed — Lost to Follow-up | 20
Not completed — Did Not Take Mifepristone or Misoprostol | 8
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Medication Abortion Patients
Number analyzed (Participants) | 506
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 27 [23 to 31]
Age, Customized [Count of Participants; unit: Participants]
  Age, Categorical: 15-19 years | 30
  Age, Categorical: 20-24 years | 144
  Age, Categorical: 25-29 years | 161
  Age, Categorical: Greater than or equal to 30 years | 171
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex/Gender data not collected
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and ethnicity: Black | 194
  Race and ethnicity: Hispanic | 88
  Race and ethnicity: White | 141
  Race and ethnicity: Multiracial/other race | 45
  Race and ethnicity: Missing data | 38
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 506
Educational level [Count of Participants; unit: Participants]
  High school or less | 170
  Some college or professional school | 206
  College or advanced degree | 112
  Missing data | 18
Parity [Count of Participants; unit: Participants]
  Nulliparous | 189
  Parous | 317
Prior abortion experience [Count of Participants; unit: Participants]
  None | 249
  Medication abortion | 149
  Procedural abortion only | 93
  Missing data | 15

OUTCOME MEASURES:

1. Primary Outcome: Acceptability: Satisfaction With Mail-Order Dispensing of Medication Abortion
Description: Percentage of participants reporting whether they were satisfied with receiving the medications by mail, by abortion instance.
Time Frame: Day 14 following initial medication abortion visit
Measure: Count of Units; unit: Number of abortions
Units Other Than Participants: Number of abortions
Arm/Group | Medication Abortion Patients
Number analyzed (Participants) | 491
Number analyzed (Number of abortions) | 495
Number of abortions
  Very satisfied | 452
  Somewhat satisfied | 26
  Neither satisfied nor dissatisfied | 7
  Somewhat dissatisfied | 4
  Very dissatisfied | 6

2. Primary Outcome: Acceptability: Would Use Mail-Order Dispensing Again
Description: Percentage of participants reporting they would prefer to receive medications by mail for future medication abortion, by abortion instance.
Time Frame: Day 14 following initial medication abortion visit
Measure: Count of Units; unit: Number of abortions
Units Other Than Participants: Number of abortions
Arm/Group | Medication Abortion Patients
Number analyzed (Participants) | 473
Number analyzed (Number of abortions) | 477
Number of abortions
  Yes | 431
  No | 20
  Not sure | 26

3. Secondary Outcome: Feasibility: Proportion of Patients Who Receive Medications by Day 2 and Day 3
Description: Percentage of participants who received the medications by mail-order pharmacy by Day 2 and Day 3, by abortion instance.
Time Frame: Day 3 following initial medication abortion visit
Measure: Count of Units; unit: Number of abortions
Units Other Than Participants: Number of abortions
Arm/Group | Medication Abortion Patients
Number analyzed (Participants) | 506
Number analyzed (Number of abortions) | 510
Number of abortions
  Medications delivered by Day 2 | 381
  Medications delivered by Day 3 | 436

4. Secondary Outcome: Feasibility: Confidentiality Maintained When Receiving Medications by Mail
Description: Percentage of participants who reported that confidentiality was maintained when they received the medications by mail-order pharmacy, by abortion instance.
Time Frame: Day 3 following initial medication abortion visit
Measure: Count of Units; unit: Number of abortions
Units Other Than Participants: Number of abortions
Arm/Group | Medication Abortion Patients
Number analyzed (Participants) | 491
Number analyzed (Number of abortions) | 495
Number of abortions
  Yes, confidentiality was maintained | 486
  No, confidentiality was compromised | 8
  Missing data | 1

5. Secondary Outcome: Clinical Effectiveness of Mail-Order Medication Abortion
Description: Percentage of participants who experienced a complete medication abortion, by abortion instance.
Time Frame: Up to 6 weeks after initial medication abortion visit.
Measure: Count of Units; unit: Number of abortions
Units Other Than Participants: Number of abortions
Arm/Group | Medication Abortion Patients
Number analyzed (Participants) | 506
Number analyzed (Number of abortions) | 510
Number of abortions
  Abortion complete with medications only | 499
  Incomplete abortion | 5
  Ongoing pregnancy | 6

6. Secondary Outcome: Clinical Safety of Mail-Order Medication Abortion
Description: Percentage of participants who experience adverse events related to the abortion, by abortion instance.
Time Frame: Up to 6 weeks after initial medication abortion visit.
Measure: Count of Units; unit: Number of abortions
Units Other Than Participants: Number of abortions
Arm/Group | Medication Abortion Patients
Number analyzed (Participants) | 506
Number analyzed (Number of abortions) | 510
Number of abortions
  Adverse Event Related to Medication Abortion | 21
  Serious Adverse Event Related to Medication Abortion | 3
  Adverse Event Related to Mail-Order Dispensing | 0

7. Secondary Outcome: Provider Acceptability of Mail-Order Dispensing of Medication Abortion
Description: Provider acceptability will be assessed qualitatively through open-ended interviews with providers and staff involved in the study.
Time Frame: Up to 3 months after data collection completed.
Population: Clinicians and staff involved in implementing a mail-order dispensing model for medication abortion were invited to complete qualitative interviews to share their experiences with non-in-person dispensing of mifepristone. These clinicians and staff were not officially enrolled as participants in the study, but rather contributed perspectives as clinic employees on the feasibility and acceptability of such a model.
Measure: Number; unit: participants
Groups:
- Staff and Clinicians Involved in Mail-order Dispensing at Study Sites: Oral Mifepristone 200 mg, followed by misoprostol 800 mcg administered buccally (at 24-48 hours following mifepristone)
  Mifepristone: Patients will have MifeprexⓇ (mifepristone) shipped to a preferred address via an online mail order pharmacy rather than standard care at clinic visit.
Arm/Group | Staff and Clinicians Involved in Mail-order Dispensing at Study Sites
Number analyzed (Participants) | 24
participants | 24

ADVERSE EVENTS:
Time Frame: Follow-up data were collected among participants up to six weeks after initial medication abortion visit.
Description: Adverse events were defined as any unscheduled visits, including emergency department visits, for symptoms possibly related to the medication abortion. Serious adverse events were defined as death, hospitalization, blood transfusion, or surgery.
Arm/Group | Medication Abortion Patients
All-Cause Mortality (participants affected / at risk) | 0/510
Serious Adverse Events (participants affected / at risk) | 3/510
Other Adverse Events (participants affected / at risk) | 21/510
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medication Abortion Patients (N=510)
Hemorrhage requiring blood transfusion (Reproductive system and breast disorders) | 1 (1)
Hospitalization (Reproductive system and breast disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medication Abortion Patients (N=510)
Bleeding (Reproductive system and breast disorders) | 9 (9)
Pain (Reproductive system and breast disorders) | 9 (9)
Nausea/vomiting (General disorders) | 3 (3)
Infection (Reproductive system and breast disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Incomplete abortion (Surgical and medical procedures) | 2 (2) — Less than 5% of medication abortion cases lead to incomplete abortions; in these cases, the patients visited the emergency department with symptoms and received aspiration procedures to complete their abortions
Dehydration (General disorders) | 1 (1)
Vaginitis (Reproductive system and breast disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Lack of randomization may limit generalizability. Clinical sites that agreed to participate had at least 1 motivated clinician and a supportive administrative environment and were located in states with relatively few abortion restrictions. Study participants were open to mail-order dispensing, but this option may not be acceptable/feasible for all patients. The study was not powered to precisely estimate safety outcomes. Satisfaction may be overestimated due to social desirability bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/04/NCT03913104/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT03913104/ICF_001.pdf